CLINICAL TRIAL: NCT03187925
Title: A Complete Title Used for Approval Letters. Cervical Diverticulum Prospective, Multi-Institutional Study Proposal
Brief Title: Cricopharyngeal Dysfunction and Esophageal Diverticulum
Status: Recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Rebecca Howell, assistant professor, University of Cincinnati
Other Study IDs: 2016-6955
Record Dates: First submitted 2017-06-02; First posted 2017-06-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Zenker Diverticulum; Progressive Dysphagia; Pharyngoesophageal Diverticulum
MeSH Terms: conditions — Zenker Diverticulum | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: open, transcervical versus rigid endoscopic treatment — The goal of the project is to perform the first prospective, multi-institutional long-term (5 year) study comparing the outcomes of open, transcervical versus rigid endoscopic treatment of cervical esophageal diverticulum and cricopharyngeal dysfunction in resolving associated symptoms, complications, and recurrence rates of dysphagia surgery. This study will also include cricopharyngeal bar as it pertains to an early Zenker's diverticulum.
  Other Names: observation

SUMMARY:
Patients undergoing open transcervical or endoscopic approach in which a laser or stapler is used to divide the common wall between the diverticulum and esophagus, or who are not surgical candidates but agree to follow-up.

DETAILED DESCRIPTION:
A prospective, multi-institutional study comparing the effectiveness of the above procedures will provide a large cohort using standardized diagnostic studies, diverticulum size measurements, treatment approaches, pre-operative and post-operative assessment of symptoms in order to both compare the effectiveness of the procedures and to stratify the patients in order to determine whether demographics such as age, pre-operative size, and/or peri-operative co-morbidities influence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cervical esophageal diverticulum, with Zenker's as most common, or CP bar (with diagnosis of early Zenker) as indicated on an esophagram who the participating institutions enroll regardless of surgical management and future treatments. Patients undergoing open transcervical or endoscopic approach in which a laser or stapler is used to divide the common wall between the diverticulum and esophagus, or who are not surgical candidates but agree to follow-up.

Exclusion Criteria:

* Patients who undergo division of the common wall between the diverticulum and esophagus using flexible endoscopy will not be included in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No intended gender or racial/ethnic distribution. Intended age range is 18-100 years of age. The vulnerable population (patients) will be protected from potential coercion or undue influence as this is an observational study with elective participation in follow-up patient surveys in which patient data will otherwise be deidentified upon inspection
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Add to the paucity of dysphagia outcomes data after surgical treatment of Zenker's diverticulum. | 5 years
  Demographic data will be summarized for categorical and continuous measures. Continuous data will be compared between groups using student's t-test.
Include dysphagia outcomes comparing both endoscopic and open repair of Zenker's diverticulum to develop preliminary evidence-based indications and long-term outcomes, exploring various relevant subset analyses. | 5 years
  Would standardize the above data and lend increased power due to its multi-institutional nature. The post-operative data will include the following surveys EAT-10, RSI, VHI in order to assess for post-operative resolution of symptoms as well as an esophagram at 12month

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Howell, MD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Health Otolaryngology-Head and Neck Surgery, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Background] Bock JM, Van Daele DJ, Gupta N, Blumin JH. Management of Zenker's diverticulum in the endoscopic age: current practice patterns. Ann Otol Rhinol Laryngol. 2011 Dec;120(12):796-806. doi: 10.1177/000348941112001205. PMID 22279951
- [Background] Leong SC, Wilkie MD, Webb CJ. Endoscopic stapling of Zenker's diverticulum: establishing national baselines for auditing clinical outcomes in the United Kingdom. Eur Arch Otorhinolaryngol. 2012 Aug;269(8):1877-84. doi: 10.1007/s00405-012-1945-3. Epub 2012 Feb 17. PMID 22350426
- [Background] Parker NP, Misono S. Carbon dioxide laser versus stapler-assisted endoscopic Zenker's diverticulotomy: a systematic review and meta-analysis. Otolaryngol Head Neck Surg. 2014 May;150(5):750-3. doi: 10.1177/0194599814521554. Epub 2014 Feb 4. PMID 24496741
- [Background] Verdonck J, Morton RP. Systematic review on treatment of Zenker's diverticulum. Eur Arch Otorhinolaryngol. 2015 Nov;272(11):3095-107. doi: 10.1007/s00405-014-3267-0. Epub 2014 Sep 7. PMID 25194579
- [Background] Wilken R, Whited C, Scher RL. Endoscopic staple diverticulostomy for Zenker's diverticulum: review of experience in 337 cases. Ann Otol Rhinol Laryngol. 2015 Jan;124(1):21-9. doi: 10.1177/0003489414542421. Epub 2014 Jul 15. PMID 25026961
- [Background] Venkatesan NN, Evangelista LM, Kuhn MA, Belafsky PC. Normal fluoroscopic appearance status post-successful endoscopic Zenker diverticulotomy. Laryngoscope. 2017 Aug;127(8):1762-1766. doi: 10.1002/lary.26446. Epub 2017 Jan 4. PMID 28052332